CLINICAL TRIAL: NCT05333978
Title: Optoacoustic Detection of Inflammation Using Multispectral Optoacoustic Tomography
Brief Title: Optoacoustic Detection of Inflammation Using MSOT Device
Acronym: OU-SCC-O-FLAME
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reasons.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OU-SCC-O-FLAME
Record Dates: First submitted 2022-02-21; First posted 2022-04-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Graft Vs Host Disease; Colitis; Crohn Disease
Keywords: Imaging device; inflammatory diseases
MeSH Terms: conditions — Graft vs Host Disease; Colitis; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Imaging of Inflammatory region (Experimental): Inflammatory regions of patients scheduled for standard of care clinical visits will be imaged using the MSOT device before and after 4 weeks of treatment.
  The temperature of their skin prior to and after MSOT imaging will also be measured.
  Interventions: Device: MSOT Device; Procedure: Temperature Measurement

INTERVENTIONS:
Device: MSOT Device — The MSOT Device will be used to take images of the areas of inflammation in patients with inflammatory diseases such as GVHD, Colitis, and IBD, prior to, and after 4 weeks of treatment.
Procedure: Temperature Measurement — The temperature of the skin will be measured prior to and after each instance of MSOT imaging.

SUMMARY:
The purpose of this study is to evaluate the safety and potential of a new experimental imaging instrument called multispectral optoacoustic tomography (MSOT) to detect inflammation in patients with chronic graft versus host disease of the skin or GI tract, Crohn's disease, or Colitis disease.

DETAILED DESCRIPTION:
This is a single arm, 3-cohort study that is designed to provide safety information regarding the use of the Acuity MSOT device in the clinical setting, and the ability of MSOT imaging data to correlate with clinical findings identified via pathology or radiology.

The device will be used to obtain images of the areas of inflammation in the above patients for investigational use only, to compare to clinical pathology and patient's medical record. Patients will go through standard care procedures prior to imaging. Medically established diagnostic procedures will be used to detect areas of inflammation associated with GVHD, Crohn's, or colitis. Images using the MSOT device will be obtained through intact skin. A second MSOT scan will be performed for all patients 4 weeks post treatment. The temperature of the patient's skin will also be measured prior to and after MSOT imaging.

MSOT imaging will be for research only and no treatment decisions will be based on the MSOT images obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients documented clinical/pathologic 1) acute or chronic colon or skin GVHD, 2) Crohn's disease, or 3) colitis
* Have acceptable hematologic status [total hemoglobin (tHb) ≥ 7.0 mg/dL]
* Patients ≥ 18 yrs of age
* Willing to comply with study procedures and be available for the duration of the study
* Patient has ability to understand and the willingness to provide a signed and dated IRB-approved informed consent document.

Exclusion Criteria:

* Patients with a tattoo over the area of inflammation
* Pregnant patients are not eligible for this trial. Eligible patients (if applicable) will be required to document the date of the first day of their last menstrual cycle, and provide a negative pregnancy test if sexually active and of childbearing potential
* Patients who are breastfeeding
* Any open wound (skin ulcerations or infections) at or near the site of imaging that would preclude MSOT imaging.
* Any febrile illness that precludes or delays participation preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events due to MSOT imaging post enrollment. | 5 minutes for an MSOT image (up to 48 hours post-image)
  Proportion of patients that experience adverse events as characterized by CTCAE v5.0 resulting from MSOT imaging. The first MSOT image will be taken post-enrollment on the study. The MSOT image will take up to 5 minutes and adverse events at the time of the image (1-5 minutes) and for up to 48 hours post the image will be reported.
Adverse Events due to MSOT imaging 4 weeks after treatment. | 5 minutes for an MSOT image (up to 48 hours post-image)
  Proportion of patients that experience adverse events as characterized by CTCAE v5.0 resulting from MSOT imaging.A second MSOT image will be taken after 4 weeks of treatment.The MSOT image will take up to 5 minutes and adverse events at the time of the image (1-5 minutes) and for up to 48 hours post the image will be reported.
Measurement of skin temperature before first MSOT image post enrollment. | 1-2 minutes before the MSOT image.
  Proportion of patients with skin temperatures measured pre-MSOT imaging with a touch thermometer as part of the safety evaluation of the MSOT device. MSOT imaging will be performed after patient enrollment on the study. A temperature measurement will be recorded by placing the touch thermometer onto the skin until a temperature appears (about 30 seconds) before the MSOT image is obtained.
Measurement of skin temperature after first MSOT image post enrollment. | 1-2 minutes after the MSOT image.
  Proportion of patients with skin temperatures measured post- MSOT imaging with a touch thermometer as part of the safety evaluation of the MSOT device. MSOT imaging will be performed after patient enrollment on the study. A temperature measurement will be recorded by placing the touch thermometer onto the skin until a temperature appears (about 30 seconds) after the MSOT image is obtained.
Measurement of skin temperature before second MSOT image post-treatment. | 1-2 minutes before the MSOT image.
  Proportion of patients with skin temperatures measured pre- MSOT imaging with a touch thermometer as part of the safety evaluation of the MSOT device. MSOT imaging will be performed 4 weeks after treatment for the inflammatory disease. A temperature measurement will be recorded by placing the touch thermometer onto the skin until a temperature appears (about 30 seconds) before the MSOT image is obtained.
Measurement of skin temperature after second MSOT image post-treatment. | 1-2 minutes after the MSOT image.
  Proportion of patients with skin temperatures measured post- MSOT imaging with a touch thermometer as part of the safety evaluation of the MSOT device. MSOT imaging will be performed 4 weeks after treatment for the inflammatory disease. A temperature measurement will be recorded by placing the touch thermometer onto the skin until a temperature appears (about 30 seconds) after the MSOT image is obtained.

SECONDARY OUTCOMES:
Comparison of MSOT images to Clinical Pathology Reports for Clinical Grading of Graft Versus Host Disease. | 6 months
  Compare clinical grading (positivity/negativity; 1-4) and pathologic severity of skin and GI GVHD with extent of disease defined by clinical grading, and compare to oxy- and deoxy-hemoglobin values using MSOT localization.
Comparison of MSOT images to Clinical Pathology Reports for severity of Crohn's disease. | 6 months
  Compare clinical grading (positivity/negativity) of Crohn's disease with severity of Crohn's, and extent of disease defined by clinical grading and compare to oxy- and deoxy-hemoglobin values using MSOT localization.
Comparison of MSOT images to Clinical Pathology Reports for severity of colitis. | 6 months
  Compare clinical grading (positivity/negativity) of colitis with severity and extent of disease defined by clinical grading, and compare to oxy- and deoxy-hemoglobin values using MSOT localization.
Comparison of Collagen deposition values from MSOT images to GVHD grade/response in Clinical Pathology Reports | 6 months
  Compare mean/median collagen deposition values obtained from MSOT across GVHD grade/response.
Comparison of Collagen deposition values from MSOT images to Crohn's grade/response in Clinical Pathology Reports | 6 months
  Compare mean/median collagen deposition values obtained from MSOT across Crohn's grade/response.
Comparison of Collagen deposition values from MSOT images to colitis grade/response in Clinical Pathology Reports | 6 months
  Compare mean/median collagen deposition values obtained from MSOT across colitis grade/response.
Comparison of oxy- and deoxy-hemoglobin values from MSOT images to various prognosis criteria collected on the study for GVHD patients at diagnosis. | 6 months
  Compare mean/median oxy- and deoxy-hemoglobin values obtained from MSOT images across MAGIC score/NIH consensus and Johns Hopkins prognosis criteria collected at diagnosis in patients with acute or chronic GVHD.
Comparison of collagen deposition values from MSOT images to various prognosis criteria collected on the study for GVHD patients at diagnosis. | 6 months
  Compare mean/median collagen deposition values obtained from MSOT images across MAGIC score/NIH consensus and Johns Hopkins prognosis criteria collected at diagnosis in patients with acute or chronic GVHD.
Comparison of oxy- and deoxy-hemoglobin values from MSOT images to various prognosis criteria collected on the study for GVHD patients 4 weeks after treatment. | 6 months
  Compare mean/median oxy- and deoxy-hemoglobin obtained from MSOT images across MAGIC score/NIH consensus and Johns Hopkins prognosis criteria collected 4 weeks after treatment in patients with acute or chronic GVHD.
Comparison of collagen deposition values from MSOT images to various prognosis criteria collected on the study for GVHD patients 4 weeks after treatment. | 6 months
  Compare mean/median collagen deposition values obtained from MSOT images across MAGIC score/NIH consensus and Johns Hopkins prognosis criteria collected 4 weeks after treatment in patients with acute or chronic GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Lacey McNally, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No